CLINICAL TRIAL: NCT06240754
Title: A Pilot Study of Enasidenib for Patients With Clonal Cytopenia of Undetermined Significance and Mutations in IDH2: A Decentralized Trial
Brief Title: Enasidenib for Patients With Clonal Cytopenia of Undetermined Significance and Mutations in IDH2A Decentralized Trial
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Bristol-Myers Squibb (Industry); Damon Runyon Cancer Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202405007
Record Dates: First submitted 2024-01-16; First posted 2024-02-05 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Clonal Cytopenia of Undetermined Significance; CCUS Clonal Cytopenia of Undetermined Significance
Keywords: Clonal Cytopenia of Undetermined Significance; CCUS; IDH2; Enasidenib
MeSH Terms: interventions — enasidenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Enasidenib (Experimental): Participants will receive enasidenib 100 mg daily for 18 cycles (each cycle is 28 days).
  Participants will continue treatment with enasidenib until confirmed progression to AML or MDS, development of unacceptable toxicity, or suspicion of disease progression, provided the patient is deriving clinical benefit, which will be determined at the discretion of the principal investigator.
  Interventions: Drug: Enasidenib

INTERVENTIONS:
Drug: Enasidenib — Provided by BMS.

SUMMARY:
Study researchers think that a drug called enasidenib may help people with clonal cytopenia of undetermined significance (CCUS) because the drug blocks the mutated IDH2 protein, which may improve blood cell counts. The purpose of this study is to find out whether enasidenib is a safe and effective treatment for CCUS.

ELIGIBILITY:
Inclusion Criteria:

* Unexplained cytopenia for at least 6 months. Cytopenia is defined as the presence of ≥1 blood count indexes below the following thresholds:

  * Hgb <10 g/dL
  * ANC <1.8 × 109/L
  * Platelets <100 × 109/L
* IDH2 gene mutation (R140 or R172), performed locally, at a frequency ≥ 2%.
* At least 18 years of age.
* ECOG performance status 0-2
* Adequate organ function as defined below:

  * AST(SGOT)/ALT(SGPT) ≤ 3.0 x IULN
  * Serum total bilirubin < 1.5 x IULN (un upper limit of bilirubin 5 mg/dL is acceptable if it can be attributed to Gilbert's syndrome or erythropoiesis)
  * Creatinine clearance > 50 mL/min by Cockcroft-Gault glomerular filtration rate estimation or serum creatinine ≤ 2 x IULN
* The effects of enasidenib on the developing human fetus are unknown. For this reason, women of childbearing potential and men must agree to use adequate contraception prior to study entry, for the duration of study participation, and for 24 months after the last dose of enasidenib. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of the study, and for 4 months after the last dose of enasidenib.
* Ability to understand and willingness to sign an IRB approved written informed consent document. Legally authorized representatives may sign and give informed consent on behalf of study participants.

Exclusion Criteria:

* Indication of hematologic disease by bone marrow biopsy within 6 months of study entry.

  * Evidence of disease progression from time of bone marrow biopsy to enrollment based on investigator review of symptoms and complete blood counts
* Active malignancy (defined as > 1 cm disease on most recent CT scan in the past 6 months).
* Currently receiving therapy for solid tumor malignancy or received within the last 6 months.
* Currently receiving any other investigational agents.
* Known dysphagia, short-gut syndrome, gastroparesis, or other conditions that limit the ingestion or gastrointestinal absorption of drugs administered orally.
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to enasidenib or other agents used in the study.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia.
* Pregnant and/or breastfeeding. Women of childbearing potential must have a negative pregnancy test within 72 hours of study entry.
* Positive direct Coombs test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-10-10 (Actual); Primary Completion 2028-01-31 (Estimated); Study Completion 2029-02-28 (Estimated)

PRIMARY OUTCOMES:
Best hematologic response | Up to 18 cycles (each cycle is 28 days) of treatment (up to approximately 17 months)
  Hematologic response to enasidenib will be evaluated according to a modified version of the IWG 2006 Criteria for Hematologic Improvement for patients with MDS on clinical trials

SECONDARY OUTCOMES:
Toxicity as measured by the number of adverse events experienced by participant | From start of treatment through 30 days after the last day of treatment (up to approximately 18 months)
  Measured by CTCAE v 5.0
Change in mutant IDH2 variant allele fraction | Baseline, day 1 of cycles 3/6/9/12/15 (each cycle is 28 days), and end of treatment (up to approximately 17 months)
  The IDH2 variant allele fraction reflects the clonal dominance in the blood. Blood samples will be drawn at various time points throughout the study to determine the IDH2 variant allele fraction. The lower the IDH2 variant allele fraction the better the outcome.
Duration of hematologic improvement | From start of treatment through completion of treatment (estimated to be 17 months)

CONTACTS AND LOCATIONS:
Overall Officials: Giulia Petrone, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article after deidentification (including text, tables, figures and appendices) will be available.
Supporting Information: Study Protocol, SAP
Time Frame: The data will be available immediately following publication with no end date.
Access Criteria: The data will be available immediately following publication with no end date. Access will be provided to anyone and for any purpose.

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu